CLINICAL TRIAL: NCT02187601
Title: Beta Study to Evaluate Functionality and Equivalence of MPBA (Multi Purpose Breath Analyzer-new Generation Exalenz Breath Analyzer) Compared to Currently Approved BreathID System in Assessment of Liver Function
Brief Title: Equivalence of New Breath AnalyzerCompared to Currently BreathID System in Assessment of Liver Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meridian Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LF-BETA-EX-0614
Record Dates: First submitted 2014-07-07; First posted 2014-07-11 (Estimated); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Chronic Liver Disease (CLD); Healthy Volunteers
Keywords: CLD

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CLD with MPBA and BID (Experimental): Chronic Liver Disease (CLD) patients of all degrees will be offered to be tested on the MPBA (multi purpose breath analyzer) and BID (BreathID) on a walk- in basis with , proving they meet inclusion/exclusion criteria.
  Interventions: Device: MPBA System; Device: BreathID
- HV with MPBA and BID (Experimental): Healthy volunteers (HV) with no known liver disease will undergo the breath test with the MPBA and the BID before and after substrate ingestion.
  Interventions: Device: MPBA System; Device: BreathID

INTERVENTIONS:
Device: MPBA System — MPBA is the new generation Multi Purpose Breath Analyzer
  Other Names: Multi Purpose Breath Analyzer; BreathID LF
Device: BreathID — BreathID is the name of the original Exalenz breath analyzer system

SUMMARY:
The aim of the study is to confirm that the new generation state of the art breath analyzer gives equivalent results to the previous model of the Exalenz breath analyzer.

DETAILED DESCRIPTION:
Healthy and chronic liver disease subjects of all grades will be tested to see that the two devices give equivalent results in both devices. Subjects will be connected to both devices at the same time and will be tested for one hour.

The breath test includes automatic baseline breath collection, 13C-Methacetin ingestion in solution and breath collection post ingestion.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years of age
2. Ability and willingness to sign the Informed Consent Form

   For patient group:
3. a. Known chronic liver disease (based on medical history)

For healthy volunteers:

3.b. No known liver disease (based on medical history)

Exclusion Criteria:

1. Gastric bypass surgery or extensive small bowel resection
2. Total parenteral nutrition
3. Pregnant or breast feeding
4. Allergy to acetaminophen and/or other related medications.
5. Documented drug-related concurrent hepatotoxicity or drug-related silent steatosis or drug-related fibrosis (e.g. amiodarone, methotrexate and tamoxifen).
6. Uncontrolled malabsorption or diarrhea
7. Placement of a transjugular intrahepatic portosystemic shunt (TIPS)
8. Subject should not have taken any of the following for at least 48 hours prior to the breath test: Acyclovir, allopurinol, carbamazepine, cimetidine, ciprofloxacin, daidzein, (herbal) disulfiram, echinacea, enoxacin, famotidine, fluvoxamine, methoxsalen, mexiletine, montelukast, norfloxacin, phenylpropanolamine, phenytoin, propafenone, rifampin, terbinafine, ticlopidine, thiabendazole, verapamil, zileuton or oral contraceptives or any medication that might interfere with Methacetin metabolism or might affect CYP 1A2
9. Subject should not have taken amiodarone within the last 30 days prior to the breath test

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-08; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
DOB Peak | One hour
  The DOB (Delta over Baseline) is measured before and after ingestion of challenging test substrate: 13C- Methacetin. The peak of the DOB is indicative of liver health.

SECONDARY OUTCOMES:
Number of subjects with adverse events related to breath test substrate | 48 hours
  Adverse events within 48 hours of the breath test will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Saleh Daher, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Assaf Harofe Medical Center, Tzrifin, Israel

IPD SHARING:
Plan to Share IPD: No